CLINICAL TRIAL: NCT00562822
Title: Arthroscopic vs. Non-surgical Treatment of Osteoarthritis of the Knee
Brief Title: Surgery Versus No Surgery for Osteoarthritis (OA) of the Knee
Acronym: MRC Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mrc123456; MCT-15227
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroscopy; Restraint, Physical

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthroscopic Surgery (Active Comparator): Arthroscopic surgery optimized with physical and medical therapy
  Interventions: Procedure: Arthroscopic surgery; Other: Physical and medical therapy
- Physical and medical therapy (Active Comparator): treatment with physical and medical therapy alone
  Interventions: Other: Physical and medical therapy

INTERVENTIONS:
Procedure: Arthroscopic surgery — Arthroscopic surgery to treat unresolved symptoms of osteoarthritis of the knee
  Arms: Arthroscopic Surgery
Other: Physical and medical therapy — Treatment with physical and medical therapy alone

SUMMARY:
The purpose of this study is to discover whether arthroscopic surgery is helpful in controlling the symptoms of osteoarthritis of the knee.

DETAILED DESCRIPTION:
Although arthroscopic surgery has been widely used for osteoarthritis of the knee, scientific evidence to support its efficacy is lacking. This study will compare optimized physical and medical therapy alone with arthroscopic treatment in addition to optimized physical and medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic or secondary osteoarthritis of the knee with Grade II to IV radiographic severity as defined by the modified Kellgren and Lawrence classification

Exclusion Criteria:

* Patients with inflammatory or post-infectious arthritis
* Those who had undergone previous arthroscopic treatment for knee osteoarthritis
* Those with isolate Grade III to IV medical compartment osteoarthritis with greater than 5 degrees of varus deformity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 1999-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Function, pain and quality of life based on the WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) scores | 2 years

SECONDARY OUTCOMES:
Health utility using the Standard Gamble Technique | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Fowler, MD, Principal Investigator — Western University, Canada; Brian G Feagan, MD, Study Chair — Western University, Canada
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Moseley JB, O'Malley K, Petersen NJ, Menke TJ, Brody BA, Kuykendall DH, Hollingsworth JC, Ashton CM, Wray NP. A controlled trial of arthroscopic surgery for osteoarthritis of the knee. N Engl J Med. 2002 Jul 11;347(2):81-8. doi: 10.1056/NEJMoa013259. PMID 12110735